CLINICAL TRIAL: NCT05836571
Title: Randomized Phase 2 Study of Cabozantinib, Ipilimumab, and Nivolumab in Patients With Soft Tissue Sarcoma
Brief Title: Testing Ipilimumab and Nivolumab Combination With or Without Cabozantinib in People >= 18 Years Old With Advanced Soft Tissue Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute LAO (Unknown)
Responsible Party: Sponsor
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-03149; NCI-2023-03149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 001704; 10556 (Other: National Cancer Institute LAO); 10556 (Other: CTEP)
Record Dates: First submitted 2023-04-25; First posted 2023-05-01 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Extraskeletal Myxoid Chondrosarcoma; Locally Advanced Leiomyosarcoma; Locally Advanced Liposarcoma; Locally Advanced Undifferentiated Pleomorphic Sarcoma; Locally Advanced Unresectable Soft Tissue Sarcoma; Metastatic Soft Tissue Sarcoma; Metastatic Undifferentiated Pleomorphic Sarcoma; Unresectable Leiomyosarcoma; Unresectable Liposarcoma; Unresectable Undifferentiated Pleomorphic Sarcoma
MeSH Terms: conditions — Sarcoma; Histiocytoma, Malignant Fibrous | interventions — Biopsy; Specimen Handling; cabozantinib; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (nivolumab, ipilimumab) (Active Comparator): Patients receive nivolumab IV over 30-60 minutes and ipilimumab IV over 60-90 minutes on day 1 of each cycle. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity for 4 cycles. Patients then receive nivolumab IV over 30 minutes on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI scans, tumor biopsies, and collection of blood and urine samples throughout the trial. Patients can crossover from Arm A to Arm B at the time of disease progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Arm B (cabozantinib, nivolumab, ipilimumab) (Experimental): Patients receive cabozantinib PO QD or QOD, nivolumab IV over 30-60 minutes on day 1, and ipilimumab IV over 60-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity for 4 cycles. Patients then receive nivolumab IV over 30 minutes on day 1 and cabozantinib PO QD or QOD of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients crossing over after ≥ 4 ipilimumab + nivolumab (Arm A) cycles will receive cabozantinib and nivolumab only on Arm B; patients that cross over after < 4 ipilimumab + nivolumab (Arm A) cycles will receive the remaining cycles of ipilimumab (totaling 4 doses) plus nivolumab in combination with cabozantinib. Patients who crossover start with the every 3 weeks cycle 1 treatment even if they will not be receiving ipilimumab. Patients also undergo CT or MRI scans, tumor biopsies, and collection of blood and urine samples throughout.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cabozantinib; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and urine sample
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib — Given PO
  Arms: Arm B (cabozantinib, nivolumab, ipilimumab)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial compares the effect of immunotherapy with ipilimumab and nivolumab alone to their combination with cabozantinib in treating patients with soft tissue sarcoma that has spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cabozantinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply and may also prevent the growth of new blood vessels that tumors need to grow. By these actions it may help slow or stop the spread of cancer cells. Adding cabozantinib to the combination of ipilimumab and nivolumab may be better in stopping or slowing the growth of tumor compared to ipilimumab and nivolumab alone in patients with advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess progression free survival (PFS) of ipilimumab + nivolumab versus (vs.) the cabozantinib + nivolumab + ipilimumab combination in patients with metastatic, or locally advanced, surgically unresectable soft tissue sarcoma (STS) using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.

SECONDARY OBJECTIVES:

I. Evaluate the response rate (complete response [CR]+partial response [PR]) of ipilimumab + nivolumab vs. the cabozantinib + nivolumab + ipilimumab combination.

II. Evaluate the response rate (CR+PR) of cabozantinib + ipilimumab + nivolumab in (crossover) patients whose disease has progressed on ipilimumab + nivolumab therapy.

III. Assess the number of tumor-infiltrating CD8+ T cells in tumor biopsies before and after treatment.

EXPLORATORY OBJECTIVES:

I. Measure tumor-infiltrating CD3+ T cells and CD68+ macrophages in biopsy specimens.

II. Evaluate genomic alterations in circulating tumor DNA (ctDNA) and their potential association with therapy response or resistance.

III. Investigate whether response is associated with genetic aberrations and/or tumor mutational burden.

IV. Analyze total MET and activated MET (p1235-MET) in biopsy specimens before and after study treatment and evaluate molecular target engagement by cabozantinib (as shown by a lower phosphorylated [p]MET/MET ratio).

V. Evaluate the objective response rate in patients treated with ipilimumab + nivolumab or the cabozantinib + nivolumab + ipilimumab combination using immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive nivolumab intravenously (IV) over 30-60 minutes and ipilimumab IV over 60-90 minutes on day 1 of each cycle. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity for 4 cycles. Patients then receive nivolumab IV over 30 minutes on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) scans, tumor biopsies, and collection of blood and urine samples throughout the trial. Patients can crossover from Arm A to Arm B at the time of disease progression.

ARM B: Patients receive cabozantinib orally (PO) once daily (QD) or every other day (QOD), nivolumab IV over 30-60 minutes on day 1, and ipilimumab IV over 60-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity for 4 cycles. Patients then receive nivolumab IV over 30 minutes on day 1 and cabozantinib PO QD or QOD of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients crossing over after ≥ 4 ipilimumab + nivolumab (Arm A) cycles will receive cabozantinib and nivolumab only on Arm B; patients that cross over after < 4 ipilimumab + nivolumab (Arm A) cycles will receive the remaining cycles of ipilimumab (totaling 4 doses) plus nivolumab in combination with cabozantinib. Patients who crossover will start with the every 3 weeks cycle 1 treatment even if they will not be receiving ipilimumab. Patients also undergo CT or MRI scans, tumor biopsies, and collection of blood and urine samples throughout the trial.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic STS, specifically undifferentiated pleomorphic sarcoma (UPS), extraskeletal myxoid chondrosarcoma (EMC), liposarcoma (LPS) or non-uterine leiomyosarcoma (LMS) that are locally advanced and surgically unresectable
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam. Disease will be measured by RECISTv1.1
* Patients with prior treatment with MET or VEGFR inhibitors are allowed. However, prior cabozantinib-treated patients will not be allowed. Prior ipilimumab in combination with nivolumab-treated patients will not be allowed
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< 1.5 x institutional ULN OR glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2
* Serum albumin >= 2.8g/dL
* Lipase < 2.0 x ULN and no radiologic or clinical evidence of pancreatitis
* Urine protein/creatinine ratio (UPCR) =< 1 mg/mg
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and have undetectable HCV viral load 12 or more weeks after treatment completion. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression >= 1 month after treatment of the brain metastases. Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first 2 cycles of therapy
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients must be willing to provide blood specimens and undergo biopsies for research purposes
* Patients with baseline blood pressure (BP) lower than 140 mmHg (systolic) and 90 mmHg (diastolic). Patients on > 2 anti-hypertensive agents will be excluded
* Human immunodeficiency virus (HIV)-infected patients on effective combination antiretroviral therapy are eligible as long as HIV is well-controlled and there is undetectable viral load within 6 months. For these patients, an HIV viral load test must be completed within 28 days prior to enrollment
* The effects of nivolumab, ipilimumab, and cabozantinib on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP (defined as any female who has experienced menarche and who has not undergone surgical sterilization [hysterectomy or bilateral oophorectomy] or who is not postmenopausal) should use an adequate method to avoid pregnancy for 5 months after the last dose of investigational drug. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at the time of enrollment and within 8 days prior to each cycle. Women must not be breastfeeding
* Men who are sexually active with women of child-bearing potential (WOCBP) must use any contraceptive method with a failure rate of less than 1% per year. Men receiving cabozantinib and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 5 months after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia, stable hyperthyroidism on replacement therapy, type-1 diabetes, well-controlled on insulin, and non-clinically significant toxicities at the discretion of the study Principal Investigator
* Patients who are receiving any other investigational agents
* Eligibility of subjects receiving any medications or substances known to affect or with the potential to affect the activity of cabozantinib will be determined following review of their cases by the Principal Investigator. Patients who are taking enzyme-inducing anticonvulsant agents are not eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib, nivolumab, or ipilimumab
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Strong CYP3A4 inducers (e.g., phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's Wort) are not allowed for this study. Because the lists of these agents are constantly changing, frequently updated lists available at http://medicine.iupui.edu/clinpharm/ddis/table.asp or other reliable resources will be consulted. Patients who need to come off CYP3A4 inhibitors/inducers should adhere to a washout period of at least 5 times the half-life of the CYP3A4 inhibitors and 14 days of CYP3A4 inducers
* Patients with any other significant condition(s) that would make this protocol unreasonably hazardous are ineligible. Patients with uncontrolled intercurrent illness or clinical evidence of an active infection at the time of enrollment are ineligible
* Pregnant women are excluded from this study because cabozantinib is a receptor kinase inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cabozantinib in combination with nivolumab and ipilimumab, breastfeeding should be discontinued if the mother is treated with cabozantinib. These potential risks may also apply to other immunotherapeutic agents (ipilimumab and nivolumab) used in this study
* Patients with any of the following within 12 weeks prior to the first dose of cabozantinib: gastrointestinal bleeding, hemoptysis or pulmonary hemorrhage, radiographic evidence of cavitating pulmonary lesion(s), evidence of tumor invasion of the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum, or anus), or any evidence of endotracheal or endobronchial tumor or encasement of any major blood vessels are ineligible
* The patient is unable to swallow tablets
* The patient has a corrected QT interval calculated by the Fridericia formula (QTcF) >= 470 ms within 28 days before enrollment
* Patients with a requirement for steroid or immunosuppressive treatment should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 30 days after completion of study treatment
  Will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. The primary analysis will be a logrank test and will be performed once 52 PFS events have been observed. For Arm A (ipilimumab + nivolumab), a within-arm interim futility analysis will be performed; if at least one partial response, complete response, or stable disease (SD) (SD with duration of at least 6 months) is observed among the first 14 patients enrolled to this arm. In addition, a single interim futility analysis (Wieand rule) will be performed at 50% information (26 PFS events).

SECONDARY OUTCOMES:
Objective response rate | Up to 30 days after completion of study treatment
  Defined as complete response or partial response by RECIST v1.1. Response rates within the two study arms will be (separately) reported and will be directly compared using a two-sample test of proportions. In addition, will report the rate of objective response to cabozantinib + ipilimumab + nivolumab triplet therapy in patients who have crossed over after their disease progressed on ipilimumab + nivolumab doublet.
Number of tumor-infiltrating CD8+ T cells | Baseline and pre-cycle 3
  Will be evaluated in tumor biopsies before and after treatment. Changes between paired samples will be interpreted as being likely treatment-induced if they exceed the sampling, biological, and technical variabilities determined for the assay. Unpaired baseline and post-treatment measurements may also be assessed for correlation with response, which will shed light on possible CD8+ T cell density or infiltration requirements that could inform future trial designs.

OTHER OUTCOMES:
Tumor-infiltrating CD3+ T cells and CD68+ macrophages | Baseline and Cycle[C] 2 Day[D] 22
  Will be evaluated in tumor biopsies. Non-parametric analyses will be used.
Genetic aberrations and/or tumor mutational burden | Up to 30 days after completion of study treatment
  Will investigate whether response is associated with genetic aberrations and/or tumor mutational burden. Non-parametric analyses will be used.
T cell receptor signaling in tumor-infiltrating T cells | Baseline and C2D22
  Will be evaluated in tumor biopsies. Non-parametric analyses will be used.
Total MET and activated MET | Baseline and C2D22
  Will be evaluated in biopsy specimens before and after study treatment. Will evaluate molecular target engagement by cabozantinib (as shown by a lower phosphorylated MET/MET ratio). Non-parametric analyses will be used.
Overall response | Up to 30 days after completion of study treatment
  Will be assessed using Immune-Modified RECIST as an exploratory endpoint, for comparison to RECIST v1.1. Non-parametric analyses will be used.

CONTACTS AND LOCATIONS:
Overall Officials: A P Chen, Principal Investigator — National Cancer Institute LAO
Locations (27):
- United States (26):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada